CLINICAL TRIAL: NCT03657537
Title: KETOCOGNITION - Effects of Ketone Bodies on Cognition in Type 2 Diabetes
Brief Title: Effects of Ketone Bodies on Cognition in Type 2 Diabetes
Acronym: KETOCOGNITION
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Psychiatric Centre Rigshospitalet (Other)
Responsible Party: Principal Investigator, Nicole Jacqueline Jensen, Clinical research assistant, Bispebjerg Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-18010656
Record Dates: First submitted 2018-08-20; First posted 2018-09-05 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Type2 Diabetes; Ketonemia; Cognitive Change
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperketonemia - Placebo (Experimental): Participants are randomly assigned to initially receive ketone infusion and then saline infusion
  Interventions: Drug: Ketone infusion; Drug: Saline infusion
- Placebo - Hyperketonemia (Experimental): Participants are randomly assigned to initially receive saline infusion and then ketone infusion
  Interventions: Drug: Ketone infusion; Drug: Saline infusion

INTERVENTIONS:
Drug: Ketone infusion — β-hydroxybutyrate is infused intravenously.
Drug: Saline infusion — saline is infused intravenously.

SUMMARY:
Diabetes negatively affects cognition and increases the risk of developing overt dementia. Decreased cerebral glucose metabolism may be contributing to this effect, thus providing a glucose substitute using ketone bodies might improve neuronal function.

In this study the investigators propose to provide quantitative results on cognitive performance during acute hyperketonemia in patients with type 2 diabetes.

DETAILED DESCRIPTION:
It has been proposed that hypometabolism in the brain contributes to the neuropathology that leads to Alzheimer's disease (AD). Additionally cognitive disturbances in patients with AD are associated with and paralleled by a decrease in cerebral glucose metabolism. This AD-like reduction in cerebral metabolism has also been associated with insulin-resistance, and may contribute to one of the links between diabetes and AD. Therefore manipulating neuro-energetics by providing a glucose substitute seems to be a means of improving neuronal function.

Here the investigators will examine the effect of ketone bodies on cognitive performance in patients with type 2 diabetes by a randomized cross-over trial. Each subject will meet for two experimental visits separated by 2-6 weeks. During the two visit days subjects will, in a randomized order, receive ketone bodies (β-hydroxybutyrate) or placebo (saline) intravenously. On both test days plasma glucose levels will be clamped. After glucose levels have been stabilized cognitive performance will be assessed by a battery of validated cognitive tests.

ELIGIBILITY:
Inclusion Criteria:

* Informed and written consent
* Clinically diagnosed type 2 diabetes mellitus for at least 3 months (diagnosed according to the criteria of the World Health Organization (WHO)).
* Normal haemoglobin ≥ 8.0 mmol/L (male) or ≥ 6.4 mmol/L (female)
* Male or female participants aged 35-70 years, both inclusive.
* Treated with diet or any antidiabetic medication except insulin and SGLT2i within the last 3 weeks.
* HbA1c ≤ 9.5 % by local laboratory analysis.
* BMI > 23 kg/m2 and < 35 kg/m2

Exclusion Criteria:

* Receipt of any investigational medicinal product within 3 months prior to screening.
* Liver disease (alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) >2 times normal values) or history of hepatobiliary disorder.
* Nephropathy (serum creatinine levels ≥ 126 μmol/L (male) or ≥ 111 μmol/L (female)).
* Cardiac problems defined as decompensated heart failure (New York Heart Association (NYHA) class III and IV) at any time and/or angina pectoris within the last 12 months and/or acute myocardial infarction at any time.
* Active or recent malignant disease.
* Treatment with drugs that cannot be paused for 12 hours.
* Repeated resting blood pressure at screening outside the range 90-150 mmHg for systolic or 50-100 mmHg for diastolic. This exclusion criterion also pertains to subjects taking antihypertensives.
* Inability to perform cognitive tests as assessed by the investigators (e.g. visual or auditory impairment).
* Known abnormalities of the central nervous system or any endocrinological (with the exception of diabetes mellitus and euthyroid goiter), haematological, neurological, psychiatric diseases or other major disorders that in the opinion of the investigator precludes compliance with the protocol, evaluation of the results or represent an unacceptable risk for the participant's safety.
* Proliferative retinopathy (funduscopy performed within 12 months before the screening is acceptable) and/or severe neuropathy.
* Current treatment with systemic drugs, which may interfere with glucose metabolism.
* Significant history of alcoholism or drug/chemical abuse as per investigator's judgement.
* Current tobacco user (smoking or nicotinic product use 3 months prior to screening).
* Severe hypoglycaemic event during the past 6 months.
* Known hypoglycaemia unawareness.
* Participants with mental incapacity or language barriers precluding adequate understanding or co-operation or who, in the opinion of the investigator or their general practitioner, should not participate in the trial.
* For females only: Pregnancy, breast-feeding status or intention of becoming pregnant during the trial.
* Any chronic disorder or severe disease that in the opinion of the investigator might endanger participant's safety or compliance with the protocol.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Cognitive composite score (global score) | When glucose levels have been stabilized for 40 minutes

SECONDARY OUTCOMES:
Symbol Digit Modalities Test (SDMT) | When glucose levels have been stabilized for 40 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Research in Endocrinology, Bispebjerg University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No